CLINICAL TRIAL: NCT06157723
Title: Economic Burden of Knee Osteoarthritis in Talavera de la Reina Health Area: a Descriptive Retrospective Observational Study Using Database
Brief Title: Economic Burden of Knee Osteoarthritis in Talavera de la Reina Health Area.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Natalia Comino Suarez, PhD, University of Castilla-La Mancha
Other Study IDs: Burden Knee Osteoarthritis
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; economic burden; Physical therapy; Retrospective; Observational
MeSH Terms: conditions — Osteoarthritis, Knee; Financial Stress | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee osteoarthritis participants: Participants who are registered in the Health system electronic database, with a clinical and radiographic diagnostic of knee osteoarthritis. Approximately a total of 400 participants will be enrolled in the study.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Data related to the knee osteoarthritis will be extracted from patients' medical records:
  The sociodemographic and clinical participants' characteristics: age, weight, height, duration of the condition, and occupational activity.
  The healthcare costs: the number of visits in primary and specialized care, diagnostic tests, surgical interventions, and emergencies at both health centers and hospitals, physical rehabilitation and number of sessions.
  Charlson Comorbidity Index (CCI). Pharmacotherapy (type of drug and dose). Work absences (temporary and permanent).
  Other Names: Observational study

SUMMARY:
This is a descriptive retrospective study of individuals affected with knee osteoarthritis. The aim of this study is to describe the sociodemographic and clinical characteristics of individuals diagnosed with knee osteoarthritis within a specific health area, as well as to assess the economic impact of this condition on the healthcare system. To achieve this, medical records will be reviewed, and the following data will be collected:

Sociodemographic and clinical participant data. Healthcare resource use. Clinical burden. Up to 400 subjects will be enrolled in the Talavera de la Reina Health Area (Toledo, Spain).

DETAILED DESCRIPTION:
This is a multicenter, observational, retrospective study focusing on individuals diagnosed with knee osteoarthritis. This study will be conducted in the Talavera de la Reina Health Area (Toledo, Spain). Participants will be identified through the codes assigned in the electronic database associated with knee osteoarthritis.

Data will be collected from the initial radiologic diagnostic moment to December 31, 2019. For each participant enrolled, data from medical records will be collected and entered onto an electronic case report form (REDCap).

The sociodemographic and clinical data related to the pathology will be collected, including age, weight, height, duration of the condition, and occupational activity.

The following data will be considered as direct healthcare costs: the number of visits in primary and specialized care, diagnostic tests, surgical interventions, and emergencies at both health centers and hospitals. In addition, pharmacotherapy, rehabilitation number of sessions, and work absences (temporary and permanent) will be registered.

For cost estimation, a prevalence-based approach and a bottom-up estimation will be employed in the monetary valuation of healthcare resources, utilizing official sources.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Diagnosed with unilateral or bilateral knee osteoarthritis according to the clinical criteria of the American College of Rheumatology.
* Radiographic imaging diagnosis based on the Kellgren & Lawrence (K-L) classification.

Exclusion Criteria:

* No available X-ray.
* Pre-existing neurological diseases before the diagnostic date (stroke, Parkinson's, multiple sclerosis, ALS).
* Connective tissue disorders (Ehlers-Danlos, Marfan). Secondary cause of osteoarthritis or severe osteoarthritis (ACL tears, severe traumas, infections, or sepsis).
* Inflammatory arthropathy (any type of arthritis).
* Genetic disorders with a higher risk of developing arthropathies (Down syndrome).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with a diagnosis of knee osteoarthritis registered in the electronic database of Talavera de la Reina Health Area, Toledo, Spain.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare resource use | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  Healthcare resource use will be collected from medical records. The data will be collected by four collaborators from the healthcare system, filling out electronic forms on REDCap.
  The health direct cost will be the following:
  The number of visits in primary and specialized care and type of health professional, number and type of surgical interventions, and number of emergencies at both health centers and hospitals.
  Type and number of diagnostic tests. Pharmacotherapy (type of drug and dose). The number of sessions of physical therapy.
Participants sociodemographic characteristics | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  Age, weight, height and work activity.
Participant clinical characteristics | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  Severity of knee osteoarthritis with the radiographic Kellgren and Lawrence classification.
  Disease progression time.

SECONDARY OUTCOMES:
Charlson Comorbidity Index (CCI) | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  Mortality proGnostic with the Charlson Comorbidity Index (CCI)
Work absences | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  Number of work absences (temporary and permanent) related with knee osteoarthritis
Physical therapy treatment | Data will be collected from from the initial radiologic diagnosis registered in the electronic database to December 31, 2019.
  To know the number of subjects who received the rehabilitation program for knee osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Qualified researchers can request access to anonymized individual patient data to the IP researcher. All requests will be evaluated as the Talavera de la Reina Ethics Commitee.